CLINICAL TRIAL: NCT02325167
Title: Short-term Existential Behavioural Therapy for Informal Caregivers of Palliative Patients: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Stifterverband für die Deutsche Wissenschaft (Unknown)
Responsible Party: Principal Investigator, Martin Fegg, PD Dr. Martin Fegg, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 545-12
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: informal caregivers; mental stress; quality of life; psychotherapeutic intervention
MeSH Terms: conditions — Depression; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBT (Experimental)
  Interventions: Behavioral: EBT
- Treatment-as-usual (Experimental)
  Interventions: Behavioral: treatment-as-usual

INTERVENTIONS:
Behavioral: EBT — participants assigned to the intervention arm will receive 2 manualised therapy sessions with focus on mindfulness and activating resources delivered by trained therapists at the Clinic of Palliative Care
  Arms: EBT
Behavioral: treatment-as-usual — participants assigned to the treatment-as-usual arm will receive 2 supportive sessions delivered by trained therapists at the Clinic of Palliative Care
  Arms: Treatment-as-usual

SUMMARY:
The purpose of the study is to test the effectiveness of a short-term manualised individual psychotherapy, called Existential Behavioural Therapy (EBT), to prevent depression in informal caregivers of palliative patients.

DETAILED DESCRIPTION:
The investigators have developed and pilot-tested a short-term manualised individual psychotherapy, called Existential Behavioural Therapy (EBT), to reduce psychological distress in informal caregivers of palliative patients. The investigators propose to conduct a two-arm randomised controlled trial (RCT) to test the effectiveness of EBT against usual care for the reduction of distress and the promotion of quality of life.

Two one-to-one manualised psychotherapeutic sessions will be compared to a treatment-as-usual control group.Treatment-as-usual includes two supportive sessions.

The design will be an unblinded RCT consisting of two conditions (EBT and Treatment-as-usual), with assessment at pre- and post-treatment and follow-ups at four weeks and six months. The trial will take place in the Clinic of Palliative Care, University of Munich (Klinik und Poliklinik für Palliativmedizin der LMU München).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* informal caregivers of palliative patients at last stage of life and during bereavement;
* fluent German language skills

Exclusion Criteria:

* psychiatric conditions such as schizophrenic disorder, psychotic disorder etc.;
* pronounced cognitive impairment e.g. delirium, dementia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  A reliable and valid 9-item measure of depression

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS; Watson et al., 1988) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  two mood scales, one that measures positive affect and the other which measures negative affect
Satisfaction with Life Scale (SWLS; Diener et al., 1985) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  a short 5-item instrument designed to measure global cognitive judgments of satisfaction with life
World Health Organisation Quality-of-Life Scale (WHOQOL-BREF; Angermeyer et al., 2000) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  an abbreviated 26-item generic Quality of Life Scale developed through the World Health Organisation measuring physical health, psychological health, social relationships, and environment
Numeric rating scale for mental stress and quality of life (NRS, range 0-10) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  a numeric scale used for the subjective measurement of mental stress and quality of life
Generalised Anxiety Disorders-7 (GAD-7; Spitzer et al., 2006) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  a 7-item self-report measure designed to screen and assess the severity of generalised anxiety disorder symptoms
Fragebogen zur Inanspruchnahme medizinischer und nicht-medizinischer Versorgungsleistungen im Alter (FIMA; Seidl et al., 2014) | Baseline; 6 months follow-up
  a german questionnaire for health-related resource use
German version of the NCCN distress-thermometer (Mehnert et al., 2005) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  a subjective measurement of distress on a 0-10 scale
General Health Questionnaire (GHQ-12, Goldberg et al., 1972) | Baseline; Post-treatment; 4 weeks follow-up; 6 months follow-up
  a 12-item self-report measure of psychological morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fegg, Dr., Principal Investigator — Klinik und Poliklinik für Palliativmedizin, Ludwig Maximilians Universität München
Locations (1):
- Ludwig Maximilians University Munich, Munich, Germany